CLINICAL TRIAL: NCT05334602
Title: The Effect of Use of Dermal Fat Graft as a Barrier Membrane in Unilateral Alveolar Cleft Grafting. (A Randomized Clinical Trial
Brief Title: The Effect of Use of Dermal Fat Graft as a Barrier Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Nabil Ahmed Khirat El Hadidi, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4.12.2022
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Unilateral Cleft Lip
Keywords: Alveolar cleft grafting

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): Dermal fat graft is added over the grafted bone in the alveolar cleft to protect the bone from resorption
  Interventions: Procedure: Addition of dermal fat graft as protection over bone graft
- control group (No Intervention): Conventional procedure of alveolar cleft grafting

INTERVENTIONS:
Procedure: Addition of dermal fat graft as protection over bone graft — A barrier membrane
  Arms: study group

SUMMARY:
a study conducted to assess the use of dermal fat graft use as barrier membrane over grafted bone

DETAILED DESCRIPTION:
The study has two group in which the study will have in addition to the conventional bone grafting addition of dermal fat graft to protect the bone. The control will have just normal graft

The results are assessed using computed tomography to assess the quality of the grafted bone.

The Chisquare test was used to asses the results significance.

ELIGIBILITY:
Inclusion Criteria:

Patients having age range of 8-14ys who performed for 2ry alveolar cleft grafting at the CCC using adipose fat graft in conjunction with ACBG Boys or girls. Unilateral or bilateral cleft alveolus. Accepts Healthy Volunteers has not been entered.

Exclusion Criteria:

Younger patients requiring 1ry grafting. Older patients requiring 3ry grafting.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of oronasal fistula | 6 months
  assessment of incidence of recurrence of oronasal fistual after the surgical procedure clinically

CONTACTS AND LOCATIONS:
Overall Officials: Marwa EL Kassaby, Study Chair — Ain Shams University
Locations (1):
- Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
RCT conducted to assess the effect of adding fat over bone graft in order to protect the bone from resorption